CLINICAL TRIAL: NCT05569330
Title: Effect of Aerosol Filtering on Infectious Diseases in Day Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Ville Vartiainen, MD, PhD, MSc, researhcer, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PK-1
Record Dates: First submitted 2022-09-28; First posted 2022-10-06 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Upper Respiratory Tract Infection; Diarrhea
MeSH Terms: conditions — Respiratory Tract Infections; Diarrhea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Other): Two of the four participating day care units are allocated in arm 1
  Interventions: Other: Air purification
- Arm 2 (Other): Two of the four participating day care units are allocated in arm 2
  Interventions: Other: Air purification

INTERVENTIONS:
Other: Air purification — Aerosol particles are removed from room air by several methods

SUMMARY:
Effect of aerosol flitration and removal on typical infectious diseases such as upper respiratory tract infectinos is studied in day care. Many filtration methods such as filters and electrical filtering are used to remove aerosol particles from room air.

ELIGIBILITY:
Inclusion Criteria:

* Subject is expected to be in the same day care unit for the duration of the study

Exclusion Criteria:

* Subject is known not to be in the same day care unit for the duration of the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Incident infections | During the study periods 11/22-4/23 and 11/23-4/24. These are identical for every subject.
  Incident infections among subjects

SECONDARY OUTCOMES:
Days absent from work | During the study periods 11/22-4/23 and 11/23-4/24. These are identical for every subject.
  Days absent from work by the parents of sick children

CONTACTS AND LOCATIONS:
Overall Officials: Ville Vartiainen, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- City of Helsinki Day care, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No